CLINICAL TRIAL: NCT07030036
Title: Screening for Cognitive Disorders in Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0058_NEUROLOGIE
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Cognitive Dysfunction; Neuropsychological Tests; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to identify cognitive problems in adults with multiple sclerosis (MS). MS can affect memory, thinking speed, and spatial skills, which may impact daily life and work. We will use simple and proven tests to check for these difficulties and see how they affect quality of life. The study will include about 60 patients followed at the neurology day hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Diagnosed with multiple sclerosis (MS) for at least 6 months according to the 2017 McDonald criteria (SFSEP)
* Receiving disease-modifying treatment and followed in the neurology day hospital of CH Gonesse

Exclusion Criteria:

- Under 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (18 years and older) diagnosed with multiple sclerosis for at least six months according to the 2017 McDonald criteria. These patients are currently receiving disease-modifying treatments and are followed at the neurology day hospital of CH Gonesse.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cognitive impairment in patients with multiple sclerosis, assessed by validated cognitive tests (CSCT, RL/RI-16, Figure de REY, HAD scale, SF-12). | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France